CLINICAL TRIAL: NCT01032057
Title: A Multi-Center Randomized Phase II Study of Induction Chemotherapy Followed by Gemcitabine or Capecitabine Based Chemoradiotherapy for Locally Advanced Non-Metastatic Pancreatic Cancer
Brief Title: Gemcitabine, Capecitabine, and Radiation Therapy in Treating Patients With Locally Advanced Pancreatic Cancer That Cannot Be Removed by Surgery
Acronym: SCALOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lisette Nixon (Other)
Responsible Party: Sponsor-Investigator, Lisette Nixon, Dr, Cardiff University
Organization: Cardiff University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000660755; WCTU-SCALOP; EUDRACT-2008-001394-15; ISRCTN-96169987; WCTU-SPON-415-07; CRUK-07/040; EU-21114
Record Dates: First submitted 2009-12-13; First posted 2009-12-15 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage II pancreatic cancer; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Gemcitabine; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gemcitabine (Active Comparator): GEMCAP induction chemotherapy (28 day cycle of IV gemcitabine 1000mg/m2 day 1, 8,15 and capecitabine 830mg/m2 bd for 21 days po) followed by gemcitabine 300mg/m2 weekly (IV) + 50.4Gy radiation over five and half weeks (1.8Gy per fraction, Monday-Friday)
  Interventions: Drug: capecitabine; Drug: gemcitabine hydrochloride; Procedure: quality-of-life assessment; Radiation: 3-dimensional conformal radiation therapy
- chemoradiotherpay with capecitabine (Active Comparator): GEMCAP induction chemotherapy (28 day cycle of IV gemcitabine 1000mg/m2 day 1, 8,15 and capecitabine 830mg/m2 bd for 21 days po), followed by capecitabine 830mg/m2 bd (po, Mon-Fri) + 50.4Gy radiation over five and half weeks (1.8Gy per fraction, Monday-Friday)
  Interventions: Drug: capecitabine; Drug: gemcitabine hydrochloride; Procedure: quality-of-life assessment; Radiation: 3-dimensional conformal radiation therapy

INTERVENTIONS:
Drug: capecitabine
Drug: gemcitabine hydrochloride
Procedure: quality-of-life assessment
Radiation: 3-dimensional conformal radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy that uses a 3-dimensional image of the tumor to help focus thin beams of radiation directly on the tumor, and giving radiation therapy in higher doses over a shorter period of time, may kill more tumor cells and have fewer side effects. It is not yet known which regimen of chemotherapy given together with radiation therapy is more effective in treating pancreatic cancer.

PURPOSE: This randomized phase II trial is comparing the side effects of two regimens of gemcitabine and capecitabine given together with radiation therapy and to see how well they work in treating patients with locally advanced pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the activity, safety, and feasibility of induction chemotherapy comprising gemcitabine and capecitabine followed by two different schedules of chemoradiotherapy comprising gemcitabine or capecitabine and radiotherapy in patients with locally advanced, nonmetastatic, unresectable pancreatic cancer.
* To determine which of the two experimental arms gives the highest generic and disease-specific aspects of health-related quality of life (HRQL) following treatment.
* To determine how HRQL varies during treatment and follow up in both arms.

OUTLINE: This is a multicenter study.

All patients receive a first induction therapy comprising gemcitabine IV on days 1, 8, and 15 and oral capecitabine twice daily on days 1-21. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity. Following the first induction therapy, patients with a WHO performance status of 0-1 who are responding or have stable disease that can be encompassed within a radically treatable radiotherapy volume are randomized to 1 of 2 treatment arms.

* Arm I:

  * Second induction therapy (weeks 13-16): Patients receive gemcitabine IV once daily on days 1, 8, and 15 and oral capecitabine twice daily on days 1-21.
  * Chemoradiotherapy (weeks 17-22): Patients receive gemcitabine IV once weekly on day 1 and undergo conformal radiotherapy 5 days a week for 5.5 weeks.
* Arm II:

  * Second induction therapy (weeks 13-16): Patients receive gemcitabine IV once daily on days 1, 8, and 15 and oral capecitabine twice daily on days 1-21.
  * Chemoradiotherapy (weeks 17-22): Patients receive oral capecitabine twice daily on days 1-5 and undergo conformal radiotherapy 5 days a week for 5.5 weeks.

Patients complete quality-of-life questionnaires QLQ-C30 and PAN26 at baseline and at 17, 23, 26, 39, and 52 weeks.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Locally advanced, nonmetastatic, inoperable, or operable (but medically unfit for surgery) disease

    * Palliative bypass procedure allowed
    * Common bile duct stenting allowed
* Primary pancreatic lesion ≤ 7 cm in diameter as measured by CT scan of the thorax and abdomen within 4 weeks prior to registration
* No recurrent cancer following definitive pancreatic surgery

PATIENT CHARACTERISTICS:

* WHO performance status (PS) 0-2
* Neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Hemoglobin ≥ 10 g/dL
* Serum bilirubin < 35 μmol/L (50 μmol/L allowed for patients who have had a recent biliary drain and whose bilirubin is descending)
* AST/ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN
* GFR > 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 weeks after completion of study therapy
* No evidence of severe uncontrolled systemic diseases including uncontrolled coronary artery disease
* No myocardial infarction or stroke within the past 6 months
* No prior malignancies within the past 5 years except for carcinoma in situ of the cervix, adequately treated basal cell skin carcinoma, or any early-stage malignancy
* No suspected DPD deficiency
* No renal abnormalities (e.g., adult polycystic kidney disease, hydronephrosis, or ipsilateral single kidney)
* Must meet the following additional criteria for randomization:

  * WHO PS 0-1
  * Loss of weight no greater than 10% of that at baseline

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior and no concurrent sorivudine or analogues
* No prior radiotherapy to the upper abdomen
* No concurrent methotrexate
* No concurrent allopurinol

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2009-07; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 39 weeks (from registration) according to RECIST criteria | Assessed 39 weeks from registration

SECONDARY OUTCOMES:
Toxicity according to NCI CTCAE v.3.0 | Assessed throughout trial treatment and follow-up
Quality of life as measured by questionnaires QLQ-C30 and PAN26 at baseline and at 17, 23, 26, 39, and 52 weeks | Assessed throughout trial treatment and follow-up
Overall survival at 52 weeks and time from registration to death by any cause | Assessed 52 weeks post registration and during NHS flagging
Objective disease response according to RECIST criteria | 39 weeks post registration
Progression-free survival (time to event) according to RECIST criteria | Assessed during NHS flagging at the end of the trial
Radiotherapy quality assurance (adherence to protocol) | Upon completion of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Somnath Mukherjee, Principal Investigator — Northampton General Hospital
Locations (26):
- United Kingdom (26):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Queen Alexandra Hospital, Cosham, England
  - Castle Hill Hospital, Cottingham, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Helen Rollason Cancer Care Centre at North Middlesex Hospital, London, England
  - Royal Free Hospital, London, England
  - Hammersmith Hospital, London, England
  - Northampton General Hospital, Northampton, England
  - Scarborough General Hospital, Scarborough, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Musgrove Park Hospital, Taunton, England
  - Ninewells Hospital, Dundee, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Perth Royal Infirmary, Perth, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - Wrexham Maelor Hospital, Wrexham, Wales
  - Edith Cavell Hospital, Peterborough

REFERENCES:
- [Result] Mukherjee S, Hurt CN, Bridgewater J, Falk S, Cummins S, Wasan H, Crosby T, Jephcott C, Roy R, Radhakrishna G, McDonald A, Ray R, Joseph G, Staffurth J, Abrams RA, Griffiths G, Maughan T. Gemcitabine-based or capecitabine-based chemoradiotherapy for locally advanced pancreatic cancer (SCALOP): a multicentre, randomised, phase 2 trial. Lancet Oncol. 2013 Apr;14(4):317-26. doi: 10.1016/S1470-2045(13)70021-4. Epub 2013 Mar 6. PMID 23474363
- [Result] Fokas E, Spezi E, Patel N, Hurt C, Nixon L, Chu KY, Staffurth J, Abrams R, Mukherjee S. Comparison of investigator-delineated gross tumour volumes and quality assurance in pancreatic cancer: Analysis of the on-trial cases for the SCALOP trial. Radiother Oncol. 2016 Aug;120(2):212-6. doi: 10.1016/j.radonc.2016.07.002. Epub 2016 Aug 3. PMID 27497804
- [Result] Fokas E, Clifford C, Spezi E, Joseph G, Branagan J, Hurt C, Nixon L, Abrams R, Staffurth J, Mukherjee S. Comparison of investigator-delineated gross tumor volumes and quality assurance in pancreatic cancer: Analysis of the pretrial benchmark case for the SCALOP trial. Radiother Oncol. 2015 Dec;117(3):432-7. doi: 10.1016/j.radonc.2015.08.026. Epub 2015 Aug 29. PMID 26328939